CLINICAL TRIAL: NCT05185804
Title: Multicenter Randomized Prospective Open-label Clinical Trial of the Safety and Efficacy of Amidine Hydrochloride (DD217) in Prevention of Thrombotic Complications in Hospitalized Patients Diagnosed With COVID-19
Brief Title: Clinical Trial of Dimolegin (DD217) in Prevention of Thrombotic Complications in Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaDiall Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: АМ217-03
Record Dates: First submitted 2021-12-29; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Venous Thromboembolism
Keywords: Dimolegin; Dioxaban; DD217; factor Xa Inhibitor; anticoagulant; therapeutic anticoagulation; thromboprophylaxis; anticoagulation; venous thromboembolism; deep venous thrombosis; arterial thromboembolism; pulmonary embolism
MeSH Terms: conditions — COVID-19; Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — (+-)-(1'R*,2'S*,6'R*)-(2-hydroxy-4,6-dimethoxyphenyl)(3'-methyl-2'-(3''-methylbut-2''-enyl)-6-phenylcyclohex-3'-enyl)methanone; Enoxaparin; enoxaparin sodium

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, prospective, open-label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DD217 (Experimental): Study drug Dimolegin - DD217, 60 mg orally, 1 time per day
  Interventions: Drug: Dimolegin
- Group Clexane (Active Comparator): Reference drug Clexane, 40 mg subcutaneously, 1 time per day
  Interventions: Drug: Clexane

INTERVENTIONS:
Drug: Dimolegin — 60 mg orally, 1 time per day
  Other Names: DD217
  Arms: Group DD217
Drug: Clexane — 40 mg subcutaneously, 1 time per day
  Other Names: Enoxaparin sodium
  Arms: Group Clexane

SUMMARY:
Study purpose was to study the safety and efficacy of Dimolegin - DD217 as a drug for prevention of thrombotic complications compared to Clexane (enoxaparin sodium) - the standard therapy currently prescribed to patients hospitalized with COVID-19.

Patients who met all inclusion criteria and no exclusion criteria were randomized into two therapy groups:

* Group 1 - test drug Dimolegin - DD217 (60 mg orally, 1 time per day);
* Group 2 - reference drug Clexane (40 mg subcutaneously, 1 time per day).

The study drugs were taken once a day until:

* the discharge from the hospital due to recovery or positive dynamics;
* or up to 30 days of the patient's stay in the hospital;
* or until the Investigator decides to discontinue the therapy for other reasons. Planned: screening of up to 450 patients, randomization: 430 (215 per group). The required number of patients is 200 per group as a result of the entire study.

DETAILED DESCRIPTION:
Study purpose:

To study the safety and efficacy of Dimolegin - DD217 as a drug for prevention of thrombotic complications compared to Clexane (enoxaparin sodium) - the standard therapy currently prescribed to patients hospitalized with COVID-19.

Study objectives:

* To study the clinical efficacy of Dimolegin - DD217 as a drug for prevention of thrombotic complications in patients hospitalized with COVID-19.
* To assess the proportion of patients with the development of thrombotic complications: deep vein thrombosis (DVT), pulmonary embolism (PE), ischemic stroke, acute mycardial infarction (AMI), arterial thrombotic complications of other localizations (thrombosis of mesenteric arteries, renal arteries, spleen, upper and lower extremities) during the study therapy (maximum - 30 days).
* To evaluate the proportion of patients transferred to the ICU due to complications of COVID-19 and the all-cause mortality rate during the study therapy (maximum - 30 days) and during the study (maximum 90± 2 days); To study the safety of use, the rate of major and clinically significant minor bleeding and possible side effects of Dimolegin - DD217 during the study therapy (maximum - 30 days).

Methodology:

Multicenter randomized prospective open-label clinical study.

Patients who met all inclusion criteria and no exclusion criteria were randomized into two therapy groups:

* Group 1 - test drug Dimolegin - DD217 (60 mg orally, 1 time per day);
* Group 2 - reference drug Clexane (40 mg subcutaneously, 1 time per day). The first dosing (or administration) of the drug was performed on day 1 (D1) (screening/randomization). Further, patients received drugs according to their distribution into groups, preferably in the morning before the end of therapy, i.e. every morning patients received either an injection of Clexane 40 mg subcutaneously once a day, or test drug Dimolegin - DD217 60 mg (6 tablets of 10 mg).

The study drugs were taken once a day until:

* the discharge from the hospital due to recovery or positive dynamics;
* or up to 30 days of the patient's stay in the hospital;
* or until the Investigator decides to discontinue the therapy for other reasons. During the study therapy, 3 face-to-face follow-up visits were envisaged: Visit 2 (D3±1), Visit 3 (D5±1), Visit 4/EOT (D7-D30).

In all groups, specific antithrombotic prophylaxis was carried out only during inpatient treatment under the supervision by Investigator. The study drugs were not dispensed to the patient.

End of therapy (EOT) visit V4 was carried out in connection with the end of therapy and discontinuation of the study drugs. After the end of therapy, patients were included in the follow-up phase. The visit V5 was conducted in the form of a remote survey in 60±2 days after the end of therapy.

Number of subjects:

Planned: screening of up to 450 patients, randomization: 430 (215 per group). The required number of patients is 200 per group as a result of the entire study.

Actually included: 401 patients were screened, 400 patients were randomized (198 to the Dimolegin - DD217 group and 202 to Clexane group), 399 patients received the study drugs (197 in the Dimolegin - DD217 group and 202 in the Clexane group).

Test drug, dose and route of administration, batch number:

Test drug: Amidine hydrochloride (DD217) Dosage form: enteric-coated tablets Active substance: N-(5-chloropyridine-2-yl)-2-[(4- methylaminophenylcarbonyl)-amino]-5-methylbenzamide hydrochloride Active substance: Amidine hydrochloride 10 mg. Dosing regimen: 60 mg (6 x 10 mg tablets) orally, once a day (preferably in the morning)

Duration of treatment and follow-up:

Duration of treatment: maximum 30 days. Duration of follow-up: 60± 2 days after the end of therapy.

Reference drug, dose and route of administration, batch number:

Reference drug: Clexane Dosage form: Solution for injection Active substance: Enoxaparin sodium

Composition (for 4000 anti-Xa IU/0.4 mL, equivalent to 40 mg/0.4 mL):

Active substance: enoxaparin sodium 40 mg Dosing regimen: 40 mg subcutaneously, once a day (preferably in the morning)

Statistical methods:

Concomitant and past diseases (history), as well as adverse events were encoded using the MedDRA classifier in the current version at the time of the analysis (version 24.0). No missing data were imputed.

Analysis of efficacy endpoints:

For the primary efficacy endpoint, the hypothesis of non-inferiority of Dimolegin - DD217 compared to Clexane was evaluated.

This one-sided hypothesis was evaluated with an overall level of statistical significance of α=5 %. Two-sided 90 % confidence intervals (CI) were calculated for the tests. The hypothesis was evaluated by comparing the lower limit of the two-sided 90 % CI with the limit of non-inferiority of Δ = 10 %.

The analysis was carried out in the per protocol set (PPS). The analysis of secondary efficacy endpoints was carried out descriptively, the proportion of patients with the corresponding event is presented. Moreover, 90 % CIs were calculated for differences in proportions in Dimolegin - DD217 Group 1 compared to Clexane Group 2.

Analysis of safety endpoints:

Analysis of the primary safety endpoint (the incidence of cumulative major and clinically significant minor bleedings during the study therapy (maximum - 30 days)) was performed descriptively by presenting the proportion of patients with the corresponding event. Moreover, 90 % CIs were calculated for differences in proportions between the Dimolegin - DD217 group and the Clexane group.

The analysis of secondary safety endpoints was carried out in the same way as described for the primary safety endpoint. All other safety endpoints are analyzed descriptively.

The safety analysis population included all patients who received at least one dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed a written consent to participate in the study
* Hospitalized patients with a diagnosis: COVID-19 coronavirus disease confirmed by laboratory testing regardless of the severity of clinical signs no later than 72 hours before screening (U07.1 - virus was identified), or COVID-19 coronavirus disease, when the infection is diagnosed clinically or epidemiologically no later than 72 hours before screening, but laboratory tests are inconclusive or unavailable (U07.2 - virus was not identified), moderate form. To be classified as a moderate form, the patient must have at least one of the following criteria: Body temperature > 38 °C; respiratory rate (RR) > 22/min; shortness of breath during physical exertion; CT (radiography) findings typical of viral lesion (minimal or average lesion volume, Grade 1-2 on CT); SpO2<95 %; serum C reactive protein (CRP) > 10 mg/L
* Males and non-pregnant females (negative pregnancy test or human chorionic gonadotropin (HCG) blood test (for females with childbearing potential)) at the age of 18 to 85 years
* Patients who are able to comply with all the requirements of the study protocol;
* Patients who agreed to use adequate methods of contraception during the entire study and for at least 7 days after the end of the study

Exclusion Criteria:

* Patients treated with anticoagulants or fibrinolytics before inclusion in the study (for example, treatment of venous thromboembolism, atrial fibrillation, the presence of a mechanical prosthetic heart valve, etc.)
* The need to prescribe anticoagulants to the patient at therapeutic doses
* Active bleeding currently or within 6 months prior to screening, high risk of bleeding
* Severe anemia
* Severe thrombocytopenia
* Congenital thrombophilia (deficiency of antithrombin III, protein C, protein S, Leiden mutation of coagulation factor V, increased level of coagulation factor VIII, mutation of prothrombin G20210A, etc.)
* Other coagulation disorders and indications when anticoagulants is impossible to use according to the Investigator
* It is necessary to monitor and to treat in the ICU
* Disease with the life expectancy of <3 months
* Surgery on the brain or spinal cord, spine, ophthalmic or major surgery or injury in the last 90 days
* Gastrointestinal tract disorders that can disrupt the absorption of the study drug (Crohn's disease, ulcerative colitis, irritable bowel syndrome, etc.)
* Acute gastric or duodenal ulcer, erosive gastritis with increased risk of bleeding
* Active liver disease (viral hepatitis B or C, cirrhosis of the liver) and biliary tract disease, with the exception of non-alcoholic steatohepatitis with normal levels of hepatic transaminases
* Nephrotic syndrome, significant kidney diseases with the nephrotic syndrome events
* Severe renal failure (creatinine clearance < 30 mL/min)
* Active cancer (excluding non-melanoma skin cancer), defined as cancer without remission or requiring active chemotherapy or additional treatments such as immunotherapy or radiation therapy
* History of HIV, lues
* History of tuberculosis
* Significant drug or alcohol abuse according to the Investigator in the history or currently
* The development of trophic disorders on the lower extremities that do not respond to medical treatment
* The blood level of platelets is below 25•109L
* Body mass index (BMI) less than 18.5 or more than 40 kg/m2. Body weight below 40 kg or above 130 kg
* Systolic blood pressure (SBP) > 180 mmHg and/or diastolic blood pressure (DBP) >110 mmHg and/or SBP < 90 mmHg and/or DBP <60 mmHg
* Hypersensitivity or contraindications to DD217 or enoxaparin sodium
* Women who are pregnant or breastfeeding
* Women planning pregnancy during a clinical trial (including women who received a positive pregnancy test result at screening or before taking the study drug);
* Women of childbearing potential (including non-sterilized surgically and in the postmenopausal period less than 2 years) who do not want or cannot use adequate methods of contraception throughout the study. Adequate methods of contraception include the use of a condom or diaphragm (barrier method) with spermicide
* Participation in another clinical trial currently or within 30 days prior to screening, use of any study drug for 30 days or 5 half-lives (which is longer) prior to screening
* Inability to read or write; unwillingness to understand and follow the procedures of Study Protocol
* Failure to comply with the regimen of treatment or procedures, which, in the opinion of the Investigator, may affect the study results or the safety of the patient and prevent the patient from further participating in the study
* Any other concomitant medical or serious mental conditions that make the patient ineligible for a clinical trial, limit the validity of the informed consent, or may affect the patient's ability to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
The frequency of DVT | 30 Days
  The frequency of DVT during the study therapy (maximum - 30 days)
The frequency of PE | 30 Days
  The frequency of PE during the study therapy (maximum - 30 days)
The frequency of ischemic stroke | 30 Days
  The frequency of ischemic stroke during the study therapy (maximum - 30 days)
The frequency of AMI | 30 Days
  The frequency of AMI during the study therapy (maximum - 30 days)
The frequency of arterial thrombotic complication | 30 Days
  The frequency of arterial thrombotic complication (thrombosis of mesenteric arteries, renal arteries, spleen, upper and lower extremities) during the study therapy (maximum - 30 days)

SECONDARY OUTCOMES:
The proportion of patients transferred to the ICU | 30 Days
  The proportion of patients transferred to the ICU due to COVID-19 complications (development of acute respiratory failure (ARF), acute respiratory distress syndrome (ARDS), sepsis, etc.) during the study therapy (maximum - 30 days)
The all-cause mortality rate | 30 Days
  The all-cause mortality rate during the study therapy (maximum - 30 days)
The all-cause mortality rate during the study | 90 Days
  The all-cause mortality rate during the study (maximum 90±2 days)
The proportion of patients who stayed in the hospital more than 30 days | 30 Days
  The proportion of patients who stayed in the hospital more than 30 days (the study therapy stops after 30 days)
The number of days the patient spent in the hospital before discharge due to recovery or positive dynamics, including outpatient follow-up before 30 days expire | 30 Days
  The number of days the patient spent in the hospital before discharge due to recovery or positive dynamics, including outpatient follow-up before 30 days expire
Recovery rate | 30 Days
  Recovery rate (body temperature < 37.2 °C; oxygen saturation (SpO2) in air > 96 %; negative laboratory tests of biological material for SARS-CoV-2 RNA)
Proportion of patients requiring high-flow oxygen therapy or noninvasive ventilation (NIV) | 30 Days
  Proportion of patients requiring high-flow oxygen therapy or NIV
Changes in the hemostasis system parameters | 30 Days
  Changes in the hemostasis system parameters over the time (APTT, international normalized ratio (INR), D-dimer, Fibrinogen)
The efficacy of drugs in patients depends on the D-dimer level at screening | 30 Days
  The efficacy of drugs in patients depends on the D-dimer level at screening

OTHER OUTCOMES:
The frequency of major and clinically significant minor bleedings | 30 Days
  The frequency of major and clinically significant minor bleedings during the study therapy (maximum - 30 days)
The total frequency of all hemorrhagic complications | 30 Days
  The total frequency of all hemorrhagic complications during the study therapy (maximum - 30 days)
The frequency of clinical signs of severe thrombocytopenia | 30 Days
  The frequency of clinical signs of severe thrombocytopenia during the study therapy (maximum - 30 days)
The frequency of treatment-emergent adverse events | 30 Days
  The frequency of treatment-emergent adverse events during the study therapy (maximum - 30 days)
The frequency of treatment-emergent serious adverse events | 30 Days
  The frequency of treatment-emergent serious adverse events during the study therapy (maximum - 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry A Napalkov, Professor, Study Chair — Department of Faculty Therapy No. 1 of the Sechenov University
Locations (6):
- Russia (6):
  - Regional budgetary healthcare institution Ivanovskaya clinical hospital named after Kuvaevs, Ivanovo
  - State Budgetary Institution of Healthcare Research Institute - Regional Clinical Hospital No. 1 named after Professor S.V. Ochapov Ministry of Health of the Krasnodar Territory, Krasnodar
  - Federal State Budgetary Educational Institution of Higher Education Ryazan State Medical University named after academician I.P. Pavlova of the Ministry of Health of the Russian Federation, Ryazan
  - State Healthcare Institution Saratov City Clinical Hospital No. 2 named after IN AND. Razumovsky, Saratov
  - St. Petersburg State Budgetary Healthcare Institution City Hospital No. 40 of Kurortny District, Sestroretsk
  - State budgetary institution of health care of the Yaroslavl region Yaroslavl Regional Clinical Hospital of War Veterans - International Center for the Problems of the Elderly Healthy Longevity, Yaroslavl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tovbin DG, Tarasov DN, Malakhov DV, Tserkovnikova NA, Aybush AV, Drozd NN. The Development of New Low-Molecular-Weight Factor Xa Inhibitors that are Potential Anticoagulants. Curr Drug Discov Technol. 2022;19(1):e010921191770. doi: 10.2174/1568009621666210224104940. PMID 33655836
- [Background] Tarasov DN, Tovbin DG, Malakhov DV, Aybush AV, Tserkovnikova NA, Savelyeva MI, Sychev DA, Drozd NN, Savchenko AY. The Development of New Factor Xa Inhibitors Based on Amide Synthesis. Curr Drug Discov Technol. 2018;15(4):335-350. doi: 10.2174/1570163815666180215114732. PMID 29468977